CLINICAL TRIAL: NCT00191893
Title: Bone Effects of Subcutaneous Teriparatide Following Discontinuation of Alendronate Treatment in Postmenopausal Women With Osteoporosis
Brief Title: Bone Effects of Teriparatide Following Alendronate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7918; B3D-VI-GHCK
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

INTERVENTIONS:
Drug: teriparatide

SUMMARY:
The purpose of this study is to assess the effect of 24 months of treatment with once daily teriparatide injection (recombinant human PTH [1-34]) 20 micrograms on bone histomorphometry and architecture. Patients will include postmenopausal, osteoporotic women who have been treated long term (at least 36 months) with alendronate, as well as postmenopausal, osteoporotic women who have never been treated for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Osteoporosis: Pretreated patients currently osteoporotic or osteopenic. Treatment-naive patients currently osteoporotic
* Pretreated patients will have had at least 36 months of treatment with alendronate Na 10 mg/day or 70 mg/week. Treatment-naive patients will have no significant osteoporosis treatment in the prior 36 months, as assessed by the investigator

Exclusion Criteria:

* History of bone metabolic diseases, Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hyperparathyroidism (uncorrected), and intestinal malabsorption.
* History of malignant neoplasms in the prior 5 years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. If malignant neoplasm was ever diagnosed, patient must presently be free of disease.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2003-09; Study Completion 2006-11

PRIMARY OUTCOMES:
conventional histomorphometric parameters (bone turnover, bone formation rate, and bone volume) and microdamage accumulation from iliac crest biopsies.

SECONDARY OUTCOMES:
BMD (DXA, Holoc Delphi A),Biochemical markers of bone metabolism,3-D bone morphology by high resolution quantitative Computed Tomography (QCT)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Graz, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Prague, Czechia

REFERENCES:
- [Derived] Paschalis EP, Krege JH, Gamsjaeger S, Eriksen EF, Burr DB, Disch DP, Stepan JJ, Fahrleitner-Pammer A, Klaushofer K, Marin F, Pavo I. Teriparatide Treatment Increases Mineral Content and Volume in Cortical and Trabecular Bone of Iliac Crest: A Comparison of Infrared Imaging With X-Ray-Based Bone Assessment Techniques. J Bone Miner Res. 2018 Dec;33(12):2230-2235. doi: 10.1002/jbmr.3565. Epub 2018 Sep 14. PMID 30102789